CLINICAL TRIAL: NCT02565979
Title: Effects of Long-term Resveratrol Supplementation on Metabolic Health
Brief Title: Long-term Resveratrol and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Diabetes Fonds (Other); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15-3-037
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Pre-diabetes
Keywords: Resveratrol; Diabetes Mellitus, Type 2; Insulin Resistance; Metabolic Diseases; Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Insulin Resistance; Metabolic Diseases; Glucose Metabolism Disorders | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol (Active Comparator): resveratrol will be given for 6 months, twice daily. One pill, which contains 75 mg of resveratrol, will be provided with lunch, and the other pill of 75 mg will be provided with dinner. So in total 150 mg/day of resveratrol will be given.
  Interventions: Dietary Supplement: resveratrol
- Placebo (Placebo Comparator): placebo will be given for 6 months, twice daily. One pill will be provided with lunch and the other pill will be provided with dinner.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: resveratrol — Resveratrol will be given for 6 months, twice daily. One pill, which contains 75 mg of resveratrol, will be provided with lunch, and the other pill, also containing 75 mg will be given with dinner. So in total a dose of 150 mg/day will be given.
  Other Names: resVida (99% trans-resveratrol)
  Arms: Resveratrol
Dietary Supplement: placebo — A placebo will given for 6 months, twice daily. One pill will be provided with lunch, and the other pill will be provided with dinner.
  Arms: Placebo

SUMMARY:
The main objective of the study is to investigate if 6 months resveratrol supplementation can improve glucose tolerance in overweight/obese individuals. As secondary objectives we want to investigate whether resting energy metabolism, intra-hepatic lipid content, physical performance, body composition and quality of life change by 6 months resveratrol supplementation in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40-70 years and postmenopausal women aged 50-70 years
* BMI: 27-35 kg/m2
* Stable dietary habits: no weight gain or loss > 5kg in the last three months
* Willingness to limit consumption of resveratrol-containing food products and willingness to refrain from using resveratrol containing supplements
* Subjects will only be included when the dependent medical doctor of this study approves participation after evaluating data obtained during screening

Exclusion Criteria:

* Uncontrolled hypertension
* HbA1c > 6.5%
* Previously diagnosed with type 2 diabetes
* Medication use known to interfere with glucose homeostasis/metabolism
* Current alcohol consumption > 20 grams alcohol/day
* Subjects who do not want to be informed about unexpected medical findings during the screening /study, or do not wish that their physician is informed, cannot participate in the study.
* Participation in another biomedical study within 1 month before the start of the intervention
* Any condition, disease or abnormal laboratory test result that, in the opinion of the Investigator, would interfere with the study outcome, affect trial participation or put the subject at undue risk

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-04; Primary Completion 2019-03 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Change in Glucose Tolerance | 2x baseline and 2x after 6 months of supplemenation
  Matsuda Index calculated from double 2-hour Oral Glucose Tolerance Test (OGTT)

SECONDARY OUTCOMES:
Change in Intra-hepatic lipid content | baseline and after 6 months of supplemenation
  Intra-hepatic lipid content measured with 1H-MRS
Change in Resting energy expenditure | baseline and after 6 months of supplemenation
  energy expenditure and substrate oxidation will be measured by an automated ventilated hood system (45 minutes) to determine whole body energy metabolism
Change in Body composition | baseline and after 6 months of supplemenation
  Body composition will be assessed by dual energy X-ray absorptimetry (DEXA) scan
Change in Blood plasma markers | Once a month for a period of 6 months
  Markers related to energy metabolism (for instance glucose, insulin, free fatty acids, cholesterol, glycerol and triglycerides) will be measured regularly
Change in Blood pressure | Once a month for a period of 6 months
  blood pressure (diastolic and systolic blood pressure and heart rate) will be measured once a month
Change in Physical performance | baseline and after 6 months of supplemenation
  Physical performance will be assessed by the following tests: the Timed Chair Stand Test; the 6-minute walk test while they wear a MOX Activity Monitor; and a dynamometer (Biodex) will be used to determine isometric and isokinetic muscle strength of the extensor and flexor muscles of the knee joint
Change in Quality of life | baseline and after 6 months of supplemenation
  Quality of life (QoL) will be tested using a 32-item questionnaire. This measure quantifies QoL on the dimensions Social, Spiritual, Emotional, Cognitive, Physical, Activities of Daily Living, and Integrated QoL
Change in Quality of sleep | baseline and after 6 months of supplemenation
  Sleep quality will be measured by the 10-item Pittsburg Sleep Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Prof. Dr., Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University and Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] de Ligt M, Bergman M, Fuentes RM, Essers H, Moonen-Kornips E, Havekes B, Schrauwen-Hinderling VB, Schrauwen P. No effect of resveratrol supplementation after 6 months on insulin sensitivity in overweight adults: a randomized trial. Am J Clin Nutr. 2020 Oct 1;112(4):1029-1038. doi: 10.1093/ajcn/nqaa125. PMID 32492138